CLINICAL TRIAL: NCT06959823
Title: Evaluation of the Effect of the Integrated Innovative Bed Apparatus Developed for the Relief of Pain and Anxiety in Pediatric Patients
Brief Title: Innovative Bed Apparatus for Pediatric Pain and Anxiety Relief
Acronym: MSPSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Evin Korkmaz, assist. prof., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSPSD-2024-01; TUBITAK-2024-003625 (Other: TUBITAK)
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Pain Management; Anxiety
Keywords: child; pain; anxiety; distraction; innovative device
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSPSD Intervention Group (Experimental): Participants received multisensory pediatric support device (MSPSD) during invasive procedures.
  Interventions: Device: Multisensory Pediatric Support Device (MSPSD)
- Standard Care Group (No Intervention): Participants received standard care without any multisensory device.

INTERVENTIONS:
Device: Multisensory Pediatric Support Device (MSPSD) — Child-friendly multisensory device providing audio-visual distraction during invasive procedures.
  Arms: MSPSD Intervention Group

SUMMARY:
Pain and anxiety are common responses in pediatric patients undergoing invasive procedures and can negatively affect both immediate care outcomes and future health-care experiences. Non-pharmacological interventions, especially those involving multisensory distraction, are increasingly used to alleviate distress. This study aimed to evaluate the effectiveness of a novel, child-friendly, multisensory support device in reducing pain and anxiety in pediatric surgical patients.

Keywords: child, pain, anxiety, distraction, pediatrics, innovative device

DETAILED DESCRIPTION:
This randomized controlled trial included 48 children aged 4-12 years who were hospitalized in the pediatric surgery unit of a tertiary hospital in Istanbul, Turkey, and who underwent an invasive procedure for the first time. Participants were randomly assigned to either the intervention (n=24) or control group (n=24) using block randomization based on age and sex. The intervention group received a Multisensory Pediatric Support Device that delivered combined audio (storybook narration), visual (lights), and animated stimuli during the procedure. The control group received standard preoperative and postoperative care. Pain and anxiety were measured using the Wong-Baker FACES Pain Rating Scale and the Children's Anxiety Meter State (CAM-S), respectively.

ELIGIBILITY:
Inclusion Criteria: Children aged 4 to 12 years.

Hospitalized in the pediatric surgery ward.

Undergoing an invasive intervention (e.g., intravenous catheter insertion, intramuscular injection, wound care) for the first time during their hospital stay.

Able to communicate and understand simple instructions.

Written informed consent obtained from legal guardians and verbal assent from the child (as appropriate to developmental level).

Exclusion Criteria:

* Children with cognitive impairments or developmental delays that prevent communication or reliable self-reporting.

Children with previous experience of invasive procedures during the current hospitalization.

Children receiving sedation or pharmacological anxiolytics before the procedure.

Children or legal guardians who refuse to provide informed consent.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Pain Score Change | Before and immediately after invasive procedure.
  Assessed by Wong-Baker FACES Pain Rating Scale (min: 0, max: 10)
Anxiety Score Change | Before and immediately after invasive procedure.
  Assessed by Children's Anxiety Meter State (CAM-S) (min: 0, max: 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be made available to qualified researchers upon reasonable request. Data requests should be directed to the principal investigator via email (dr.evinkorkmaz@gmail.com). Data will be shared after publication, with a data use agreement.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting documents will be available within 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers upon submission of a research proposal and approval by the principal investigator. A data use agreement is required prior to data sharing. Data will be transferred via secure electronic methods.
URL: https://clinicaltrials.gov/

REFERENCES:
- [Background] Uman LS, Birnie KA, Noel M, Parker JA, Chambers CT, McGrath PJ, Kisely SR. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD005179. doi: 10.1002/14651858.CD005179.pub3. PMID 24108531